CLINICAL TRIAL: NCT06306859
Title: Design and Development of Health Monitoring System on Quality of Life, Self-management and Self-efficacy Among Patients Undergoing Hemodialysis
Brief Title: Development of Health Monitoring System on Patient's Well Being in Dialysis Context
Acronym: SIKIDI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Muhammadiyah Yogyakarta (Other)
Collaborators: Ministry of Education Culture, Research and Technology (Unknown)
Responsible Party: Principal Investigator, Erna Rochmawati, Dr, Universitas Muhammadiyah Yogyakarta
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SIKIDI 2024
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Quality of Life; Self Efficacy; Chronic Kidney Diseases; M-health
Keywords: Quality of life; self efficacy; chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The intervention group will be given access to m-health to monitor and education provision for about four weeks
Who Masked: Participant
Masking Description: The sample will be divided based on the schedule of hemodialysis. Intervention group will be chosen from Monday-Thursday.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SIKIDI group (Experimental): The experimental arm will be given to access to m-health to monitor and education provision.
  Interventions: Behavioral: Using m-health for monitoring and education provision
- Comparator (Active Comparator): The comparator group will be given standard care
  Interventions: Other: Standard care

INTERVENTIONS:
Behavioral: Using m-health for monitoring and education provision — The intervention group will be given access to m-health. The m-health aims to monitor patient's status i.e blood pressure, heart rate, fluid intake, dietary intake. In addition, there will be education provided through the m-health. The education will be on fluid and diet adherence
  Arms: SIKIDI group
Other: Standard care — The comparator group will be given standard and routine care
  Arms: Comparator

SUMMARY:
One of the goals in the Sustainable Development Goals (SDGs) is the availability of a healthy and prosperous life for all ages. This goal mentions health priorities i.e. non-communicable diseases. Chronic kidney failure (CRF) is one of the non-communicable diseases that is the main cause of death and disability both in the world and in Indonesia. The prevalence of CRF in Indonesia is 0.5% with 83.2% of patients being of productive age and the highest number of CRF patients in North Kalimantan, Southeast Sulawesi, DKI Jakarta and Yogyakarta. Monitoring and evaluation of patients with CRF is currently mostly carried out conventionally not using health technology that is integrated with hospital information systems. This study aims to design and provide a health information system for patients with CRF, hereinafter referred to as SIKIDI, which integrates mobile-health applications used independently by patients with existing information systems in hospitals.

DETAILED DESCRIPTION:
One of the goals in the Sustainable Development Goals (SDGs) is the availability of a healthy and prosperous life for all ages. This goal mentions health priorities i.e. non-communicable diseases. Chronic kidney failure (CRF) is one of the non-communicable diseases that is the main cause of death and disability both in the world and in Indonesia. The prevalence of CRF in Indonesia is 0.5% with 83.2% of patients being of productive age and the highest number of CRF patients in North Kalimantan, Southeast Sulawesi, DKI Jakarta and Yogyakarta. Monitoring and evaluation of patients with CRF is currently mostly carried out conventionally not using health technology that is integrated with hospital information systems. This study aims to design and provide a health information system for patients with CRF, hereinafter referred to as SIKIDI, which integrates mobile-health applications used independently by patients with existing information systems in hospitals.

This research is a multicenter basic research in four provinces. In the first year, the level of readiness and patient needs in using the mobile-health application will be seen. Furthermore, SIKIDI will be developed for monitoring the condition of patients integrated with existing systems in hospitals, and will be tested on patients with CRF at partner hospitals in DIY provinces. In addition, the ease and comfort of patients when using SIKIDI will also be seen. The output of the first year is publication in accredited national journals and prototypes of SIKIDI version 1.

In the second phase, SIKIDI version 2 will be developed which is equipped with educational features that are expected to increase patient knowledge in self-management. The trial process will be carried out at partner hospitals to see the effectiveness of educational features with patient self-management capabilities. The advantages of SIKIDI are: (1) integrated with hospital information systems; (2) include patients and families in condition monitoring; (3) improve the self-efficacy ability of patients and families. The output of year 2 is publication in reputable international journals and prototypes of SIKIDI version 2.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* has been undergoing hemodialysis >3 months
* has smartphone

Exclusion Criteria:

* emergency hemodialysis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of Life that will be measured using KDQOL before and after intervention | four weeks
  The quality of life will be measured using Kidney Disease Quality of Life, (KDQOL) before and after the intervention. The max score is 100 and minimum score is 50

SECONDARY OUTCOMES:
Self-efficacy that will be measured using CKD SE before and after | four weeks
  The self-efficacy will be measured using validated tool CKD Self-Efficaccy (CKD SE). The maximum score is 100, and the minimum score is 0

CONTACTS AND LOCATIONS:
Locations (1):
- RS PKU Muhammadiyah Bantul, Bantul, Yogy, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided
The data will be provided upon request